CLINICAL TRIAL: NCT05330156
Title: Transurethral Resection Versus Transurethral Enucleation of the Prostate: Prospective Randomized Study
Acronym: Prostate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHMED FARAHAT HASSAN, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TURP
Record Dates: First submitted 2022-03-28; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: BPH
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transurethral resection of the prostate group (TURP). (Active Comparator): the 1st group of patients will undergone Transurethral resection of the prostate for treatment of BPH
  Interventions: Procedure: Transurethral resection of the prostate
- transurethral enucleation of prostate group (TUEP) (Active Comparator): the 2nd group of patients will undergone Transurethral enucleation of the prostate for treatment of BPH
  Interventions: Procedure: transurethral enucleation of prostate

INTERVENTIONS:
Procedure: Transurethral resection of the prostate — - After an initial cysto-urethroscopy assessment done, Transurethral resection of the prostate is performed using the bipolar system with normal saline irrigation, under spinal or general anesthesia.
  Arms: Transurethral resection of the prostate group (TURP).
Procedure: transurethral enucleation of prostate — After an initial cysto-urethroscopy assessment done, transurethral enucleation of prostate is performed using the bipolar system with normal saline irrigation, under spinal or general anesthesia.
  Arms: transurethral enucleation of prostate group (TUEP)

SUMMARY:
TUERP technique could be used in prostates of all sizes with the same safety and efficacy "size independent procedure" . TUERP could be performed using the bipolar system only ,with or without the use of morcellator.

DETAILED DESCRIPTION:
Transurethral resection of the prostate (TURP) was first done in the 1920s. Since then, TURP has been considered as the gold standard treatment for BPH . However, its relatively high complication rate and postoperative recurrence necessitates further modification in the surgery technique .The resected adenomas have been reported to recur in up to 15% of cases that need a repeat surgical intervention, even by experienced surgeons in high-volume centers .

Before the era of TURP, simple open prostatectomy was the mainstay of surgical therapy. However, open simple prostatectomy has high risk of considerable intraoperative bleeding requiring transfusion. The lower abdominal incision done in open prostatectomy may result in significant postoperative pain, an extended recovery period and longer hospital stay, with greater morbidity and a perioperative mortality rate of 0.2%. In addition, TURP for large prostatic adenomas causes significantly much more bleeding with clot retention as compared to simple open prostatectomy, it also need a longer operative time, which leads to increased risk of TUR syndrome with subsequent morbidity . A new technique in which transurethral enucleation and resection of the prostate (TUERP) was developed and adopted to replicate the open enucleation of prostatic adenomas in an endoscopic way. This will combine the benefits of complete prostate enucleation in a minimally invasive technique . prostate enucleation by laser currently used as minimally invasive and save alternative to TURP, but still has not been widely accepted for some reasons, including high cost and prolonged learning curve.

TUERP technique could be used in prostates of all sizes with the same safety and efficacy "size independent procedure" . TUERP could be performed using the bipolar system only ,with or without the use of morcellator

ELIGIBILITY:
Inclusion Criteria:

* -Patients aging from 50 to 80 years old who are diagnosed with clinical symptomatic BPH.
* The patients have clear indi¬cation for endoscopic surgery (according to the guidelines).
* Clinically fit patients for surgery.
* Signed an informed consent.

Exclusion Criteria:

* Prostate cancer Previous urethral or prostate surgery Neurogenic bladder Urethral stricture Poor general condition of the patient

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — BPH disease is a male disease
Enrollment: 58 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Time of operation | intraoperative (from the start of resection or enucleation till the fixation of urethral catheter)
  time used for resection or enucleation and resection of the prostate

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED F ABBAS, MD, Principal Investigator — AUH
Locations (1):
- assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mostafa MM, Ibrahim AF, Moeen AM, Elgammal MA, El-Azab AS, Faragallah MA. Bipolar resection versus enucleation of the prostate in management of benign prostatic hyperplasia patients with large-sized prostates: a prospective randomized controlled clinical trial. BMC Urol. 2026 Jan 24. doi: 10.1186/s12894-025-02004-1. Online ahead of print. PMID 41580733